## SAMPLE OF PATIENT INFORMED CONSENT FORM \*

#### NAME OF THE RESEARCH

INVESTIGATION OF THE EFFECTS OF PROPRIOCEPTIVE NEUROMUSCULAR FACILITATION AND KINESIOLOGICAL TAPE APPLICATIONS ON HAND FUNCTIONS IN PATIENTS WITH HEMIPLEGIC STROKE WITHIN THE SCOPE OF THE INTERNATIONAL CLASSIFICATION OF FUNCTIONALITY, DISABILITY AND HEALTH (ICF)

01.01.2025

Volunteer Initials <<....>>

You are being asked to take part in a research study. Before you decide whether you want to participate, you must understand why the research is being done, how your information will be used, what the study involves, and the possible benefits, risks, and concerns you may experience. Please take the time to read the following information carefully.

### DO I HAVE TO PARTICIPATE IN THIS STUDY?

The decision to participate in the study or not is entirely yours. If you decide to participate in the study, you will be given this Informed Consent Form to sign. If you decide to participate, you can withdraw from the study anytime. This will not affect the standard of care you receive. Your physician/GP will be informed of your participation in this clinical study if you wish. You will also be removed from the study if the sponsor company decides to terminate the study.

## WHAT IS THE SUBJECT AND PURPOSE OF THE STUDY? Explain

The subject of the study is to evaluate the effects of PNF and kinesiology taping applications on hand functions in hemiplegic stroke individuals within the scope of ICF.

### **WORKING PROCEDURES:**

Within this study's scope, upper extremity evaluations will be made. Then, the study participants will be randomly divided into groups, and different treatments will be applied to each group. The treatments to be applied within this study's scope will not negatively affect the ongoing conventional physical therapy applications and will contribute more. A manual application called PNF with facilitation, re-teaching, and stimulating effect will be applied to one of the groups. The kinesiology tape's elastic stimulating and facilitating effect will be applied to the second group. Both applications will be applied to the third group.

### WHAT SHOULD I DO?

You need to attend the practices regularly and participate in the evaluation sessions before and after treatment.

## WHAT ARE THE POSSIBLE SIDE EFFECTS, RISKS, AND DISCOMFORTS OF PARTICIPATING IN THE STUDY?

The survey will not cause any harm to you or your health.

## WHAT ARE THE POSSIBLE BENEFITS OF PARTICIPATING IN THE STUDY? (Explain if any)The survey will not cause any harm to you or your health.

With your participation in the study, the possible benefits of PNF and Kinesiology taping applications and conventional physical therapy applications will be revealed in treating hemiplegic stroke. They will be included in the training programs for your treatment and the treatment of patients to be treated in the future.

## **VOLUNTARY PARTICIPATION**

I make my decision to participate in this study entirely voluntarily. I am aware that I can refuse to participate in this study or leave at any time after participation, without affecting the care and treatments I will receive at this treatment institution, and without taking any responsibility.

## WHAT IS THE COST OF PARTICIPATING IN THE STUDY?

You will not be paid or asked for money for your participation in the study.

## HOW WILL MY PERSONAL INFORMATION BE USED?

Your name and personal information will not be used at any stage, including the conduct and publication of the study.

The study sponsor company may share your study data with other companies in its group, institutions from which service is received, contracted companies, and other research organizations that will use it only for the abovementioned purposes. The study results may be published in medical publications, but your identity will not be disclosed in these publications.

If you withdraw your consent, your study data will no longer be used or shared with other people. By signing this form, I consent to using your study data as described in this form

## PEOPLE WHO CAN BE REACHED 24 HOURS DURING THE RESEARCH:

Elif ÖNDER

Tel: 0545 377 62 07

Doç.Dr.Mahmut YARAN Ondokuz Mayıs University -Faculty of Health Sciences Department of Orthotics and Prosthetics

# <u>SITUATIONS THAT WILL REQUIRE ME TO LEAVE THE STUDY: If any, please explain</u>

If you do not agree to participate in the study or if you withdraw from the study for any reason, the care and treatments you will receive at this treatment institution will not be affected and there will be no disruption.

### **HOW MAY NEW INFORMATION AFFECT MY ROLE IN THE STUDY**

All new information that emerges during the study will be communicated to me immediately.

Consent to Participate in the Study

I have read all the explanations in the Informed Consent Form. The written and verbal explanation regarding the research whose subject and purpose are specified above was made to me by the physician named below. I know that I am participating in the study voluntarily, that I can withdraw from the study at any time with or without justification, and that I can be excluded from the study by the researcher regardless of my own will.

I agree to participate in the study of my own free will, without any pressure or coercion. A copy of this document, including the points I will pay attention to during the study, has been delivered to me for safekeeping.

Volunteer Name / Surname / Signature / Date

Person Making the Statements Name / Surname / Signature / Date

If Necessary, Person Witnessing the Consent Process Name / Surname / Signature / Date

If Necessary, Legal Representative Name / Surname / Signature / Date